CLINICAL TRIAL: NCT02063100
Title: Efficacy and Safety of Shenyankangfu Tablets for Primary Glomerulonephritis-a Multicentre, Prospective, Double-blind, Double-dummy, Randomized Controlled Clinical Trial
Brief Title: Efficacy and Safety of Shenyankangfu Tablets for Primary Glomerulonephritis
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chinese PLA General Hospital (Other)
Collaborators: Tianjin TongRenTang Group Co., Ltd. (Unknown)
Responsible Party: Principal Investigator, Chen Xiangmei, Professor, Chinese PLA General Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: S2013-055-03
Record Dates: First submitted 2014-02-12; First posted 2014-02-14 (Estimated); Last update posted 2015-07-01 (Estimated); Status verified 2015-06

CONDITIONS: Glomerulonephritis; Proteinuria
Keywords: Glomerulonephritis; proteinuria; shenyankangfu tablets; Losartan Potassium; efficacy; safety
MeSH Terms: conditions — Glomerulonephritis; Proteinuria | interventions — Losartan

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- Shenyankangfu tablets and Losartan potassium 100mg (Experimental)
  Interventions: Drug: Shenyankangfu tablets and Losartan potassium 100mg
- Shenyankangfu tablets and Losartan potassium 50mg (Experimental)
  Interventions: Drug: Shenyankangfu tablets and Losartan potassium 50mg
- Losartan potassium 50mg (Experimental)
  Interventions: Drug: Losartan potassium 50mg
- Shenyankangfu tablets (Experimental)
  Interventions: Drug: Shenyankangfu tablets
- Losartan potassium 100mg (Experimental)
  Interventions: Drug: Losartan potassium 100mg

INTERVENTIONS:
Drug: Shenyankangfu tablets — Shenyankangfu tablets 2.4g, po, 3/day and Losartan potassium placebo 2 tab, po, 1/day,all drugs and placebo are taken for 48 weeks.
  Arms: Shenyankangfu tablets
Drug: Losartan potassium 50mg — Shenyankangfu tablets placebo 5 tab, po, 3/day and losartan potassium 50mg,po, 1/day and losartan potassium placebo1 tab,po, 1/day, all drugs and placebo are taken for 48 weeks.
  Arms: Losartan potassium 50mg
Drug: Shenyankangfu tablets and Losartan potassium 50mg — Shenyankangfu tablets 2.4g, po, 3/day and losartan potassium 50mg,po, 1/day and losartan potassium placebo1 tab, po, 1/day, all drugs and placebo are taken for 48 weeks.
  Arms: Shenyankangfu tablets and Losartan potassium 50mg
Drug: Shenyankangfu tablets and Losartan potassium 100mg — Shenyankangfu tablets 2.4g, po, 3/day and losartan potassium 50mg×2,po, 1/day, all drugs and placebo are taken for 48 weeks.
  Arms: Shenyankangfu tablets and Losartan potassium 100mg
Drug: Losartan potassium 100mg — Shenyankangfu tablets placebo 5 tab, po, 3/day and losartan potassium 50mg×2,po, 1/day, all drugs and placebo are taken for 48 weeks.
  Arms: Losartan potassium 100mg

SUMMARY:
-Evaluate the efficacy and safety of Shenyankangfu Tablets to control the proteinuria of patients with primary glomerulonephritis compare with Losartan potassium.

ELIGIBILITY:
Inclusion

* Diagnosed with primary glomerulonephritis
* Aged from 18 to 70 years，male or female
* Blood pressure can be controlled ≤140/90mmHg
* GFR≥45ml/min/1.73㎡
* 0.5g≤24 hours proteinuria≤3.0g
* Traditional Chinese medicine syndrome conform Qi-Yin Deficiency
* Obtain the agreement of patients or their guardians, and signed informed consent file

Exclusion Criteria:

* secondary nephropathy
* Take the glucocorticoid,immunosuppressants and Tripterygium drug in the last 12 months
* Take other Chinese patent medicine and decoction which can reduce proteinuria in the last 2 weeks
* Take renin-angiotensin system blockers in last 4 weeks
* Combined with severe primary disease of heart, brain, liver and hematopoietic system, or other serious diseases can affect patient's life
* Pregnant or lactating women
* Allergic predisposition or known to be allergic to the drug composition
* Blood presser <90/60mmHg
* With unilateral or bilateral renal artery stenosis
* With mental disorders and poor compliance
* Be suspected or confirmed with alcohol, drug abuse history
* Be participating in another clinical study at the same period

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 720 (Estimated)
Dates: Start 2014-02; Primary Completion 2015-07 (Estimated)

PRIMARY OUTCOMES:
changes of 24 hours proteinuria after the treatment | 0,4,8,12,24,36,48 weeks after the enrollment

SECONDARY OUTCOMES:
changes of serum creatinine after treatment | 0,4,8,12,24,36,48 weeks after the enrollment
changes of eGFR after the treatment | 0,4,8,12,24,36,48 weeks after the enrollment
changes of Traditional Chinese Medicine syndrome scores after the treatment | 0,4,8,12,24,36,48 weeks after the enrollment

CONTACTS AND LOCATIONS:
Overall Officials: xiangmei chen, Doctor, Principal Investigator — State Key Laboratory of Kidney Diseases,Chinese PLA General Hospital
Locations (43):
- China (43):
  - National Clinical Research Center for Kidney Disease, State Key Laboratory of Kidney Disease, Department of Nephrology, Chinese PLA General Hospital, Beijing, Beijing Municipality
  - Beijing Friendship,Capital Medical University, Beijing, Beijing Municipality
  - Guang'anmen Hospital, China Academy of Chinese Medical Sciences, Beijing, Beijing Municipality
  - XIyuan Hospital CACMS, Beijing, Beijing Municipality
  - Daping Hospital,Research Institute of Surgery Third Military Medical University, Chongqing, Chongqing Municipality
  - Fuzhou General Hospital Nanjing Military Command, Fuzhou, Fujian
  - 174th hospital of the People's Liberation Army, Xiamen, Fujian
  - Guangdong Province Hospital of Chinese Medical, Guangzhou, Guangdong
  - Guangzhou First People's Hospital, Guangzhou, Guangdong
  - Beidaihe Sanatorium of Beijing Military Mrca, Qinhuangdao, Hebei
  - The Third Hospital of hebei Medical University, Shijiazhuang, Hebei
  - Heilongjiang University of Chinese Medicine, Harbin, Heilongjiang
  - Henan Provincial People'S Hospital, Zhengzhou, Henan
  - The Second Xiangya Hospital of Central South University, Changsha, Hunan
  - The Third Xiangya Hospital of Central South University, Changsha, Hunan
  - Xiangya Hospital Central South University, Changsha, Hunan
  - Jiangsu Province Hospital, Nanjing, Jiangsu
  - Jiangxi Provincil People'S Hospital, Nanchang, Jiangxi
  - The Second Hospital of Jilin University, Changchun, Jilin
  - First Affilated Hospital of Dalian Medical University, Dalian, Liaoning
  - Shaanxi Traditional Chinese Medicine Hospital, Xi'an, Shaanxi
  - Tangdu Hospital, Xi'an, Shaanxi
  - The First Affiliated Hospital of Xi'An Jiaotong University, Xi'an, Shaanxi
  - Xijing Hospital, Xi'an, Shaanxi
  - Shandong Province Hospital, Jinan, Shandong
  - Teaching Hospital of Shandong University of Traditional Chinese Medicine, Jinan, Shandong
  - Changhai Hospital of Shanghai, Shanghai, Shanghai Municipality
  - LONGHUA Hospital Shanghai University of TCM, Shanghai, Shanghai Municipality
  - Shanghai Jiao Tong University School of Medicine, Shanghai, Shanghai Municipality
  - Shanghai Sixth People's Hospital Affiliated to Shanghai JiaoTong University, Shanghai, Shanghai Municipality
  - Shugaung Hospital, Shanghai, Shanghai Municipality
  - Xin Hua Hospital Affiated to Shanghai Jiao Tong University School of Medicine, Shanghai, Shanghai Municipality
  - First Hospital of Shanxi Medical University, Taiyuan, Shanxi
  - Second Hospital of Shanxi Medical University, Taiyuan, Shanxi
  - Shanxi Hospital of Integrated Traditional and Westem Medicine, Taiyuan, Shanxi
  - Shanxi Provincial People's Hospital, Taiyuan, Shanxi
  - General Hospital of Chengdu Military Region of PLA, Chengdu, Sichuan
  - Teaching Hospital of Chengdu University of T.C.M, Chengdu, Sichuan
  - First Teaching Hospital of Tianjin University of TCM, Tianjin, Tianjin Municipality
  - Tianjin Medical University General Hospital, Tianjin, Tianjin Municipality
  - Hangzhou Hospital of Traditional Chinese Medicine, Hangzhou, Zhejiang
  - Tongde Hospital of Zhejiang Province, Hangzhou, Zhejiang
  - Zhejiang Provncial People'S Hospital, Hangzhou, Zhejiang

REFERENCES:
- [Derived] Wu J, Duan SW, Yang HT, Deng YY, Li W, He YN, Ni ZH, Zhan YL, Lin S, Guo ZY, Zhu J, Fang JA, Liu XS, Wang LH, Wang R, Wang NS, Cheng XH, He LQ, Luo P, Sun SR, Sun JF, Yin AP, Jiang GR, Chen HY, Liu WH, Lin HL, Liang M, Ma L, Chen M, Song LQ, Chen J, Zhu Q, Xing CY, Li Y, Gao JN, Li RS, Li Y, Zhang H, Lu Y, Zhou QL, Fu JZ, He Q, Cai GY, Chen XM. Efficacy and safety of Shenyankangfu Tablet, a Chinese patent medicine, for primary glomerulonephritis: A multicenter randomized controlled trial. J Integr Med. 2021 Mar;19(2):111-119. doi: 10.1016/j.joim.2021.01.009. Epub 2021 Jan 30. PMID 33589406
- [Derived] Kou J, Wu J, Yang HT, He YN, Fang JA, Deng YY, Xie YS, Nie LF, Lin HL, Cai GY, Chen XM. Efficacy and safety of Shenyankangfu tablets for primary glomerulonephritis: study protocol for a randomized controlled trial. Trials. 2014 Dec 5;15:479. doi: 10.1186/1745-6215-15-479. PMID 25480673